CLINICAL TRIAL: NCT05712135
Title: Investigation of Endotracheal Cuff Pressure Changes According to Different Positions in Neurosurgery Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, sena sarıcaoğlu, assistant doctor, Ankara City Hospital Bilkent
Other Study IDs: E2-22-1369
Record Dates: First submitted 2022-11-27; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: The Effect of Cuff Pressure on Postoperative Dysphagia
Keywords: cuff pressure; postoperative dysphagia; different positions in neurosurgery
MeSH Terms: interventions — Supine Position; Prone Position

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- supine: The patient group whose cuff pressure was measured in the supine position in neurosurgery
  Interventions: Other: supine position
- prone: The patient group whose cuff pressure was measured in the prone position in neurosurgery
  Interventions: Other: prone position
- semi-fowler: The patient group whose cuff pressure was measured in the semi-fowler position in neurosurgery
  Interventions: Other: semi-fowler position

INTERVENTIONS:
Other: supine position — The patient group whose cuff pressure was measured in the supine position
  Groups: supine
Other: prone position — The patient group whose cuff pressure was measured in the prone position
  Groups: prone
Other: semi-fowler position — The patient group whose cuff pressure was measured in the semi-fowler position
  Groups: semi-fowler

SUMMARY:
We aimed to measure the change in cuff pressure in different positions in neurosurgery cases and to investigate the effect of case length on cuff pressure.

DETAILED DESCRIPTION:
It is an observational study, the cuffs of the endotracheal tubes of the patients who were intubated under general anesthesia between February 2023 and May 2023 will be inflated at 25 cm H2O pressure, and then the pressure line and the pilot balloon will be connected to the anesthesia monitor. The cuff pressure of the patient will be measured from the pilot balloon throughout the case and recorded at half-hour intervals. Postoperative sore throat will be evaluated on the VAS scale. Postoperative cough, hoarseness, and dysphagia symptoms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgery patients between the ages of 18-70 ages
* American Society of Anesthesiologist score I-II-III-IV

Exclusion Criteria:

* Patients with previous tracheostomy
* Patients with tracheal stenosis
* Patients considered as difficult intubation
* Patients who have had more than one intubation attempt
* Patients with an ASA score greater than 4
* Patient who has difficulty understanding visual analog scale (VAS) scores
* Language / communication barrier
* Patients younger than 18 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgery patients between the ages of 18-70 under general anesthesia in the operating room between February 2022 and April 2022.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-05-02 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
The effect of cuff pressure on postoperative sore throat | 24 hours
  The primary outcome of the study was intubated under general anesthesia, endotracheal cuff of patients in supine, prone, semi-fowler position is to observe the change of pressures according to the positions.

SECONDARY OUTCOMES:
Comparison of cuff pressure changes with cuff time according to groups | 8 hours
  Secondary outcome of the study, case length on endotracheal cuff pressure is to observe.

IPD SHARING:
Plan to Share IPD: No